CLINICAL TRIAL: NCT06826430
Title: A Multi-center, Open-label, Single-arm Phase I Clinical Study to Evaluate the Safety and Tolerability of Inaticabtagene Autoleucel Injection in Treatment of Refractory Systemic Lupus Erythematosus-related Immune Thrombocytopenia
Brief Title: Inaticabtagene Autoleucel Injection in the Treatment of Refractory Systemic Lupus Erythematosus-related Immune Thrombocytopenia
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Juventas Cell Therapy Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HY001105
Record Dates: First submitted 2025-02-06; First posted 2025-02-14 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-08

CONDITIONS: Autoimmune Thrombocytopenia
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single dose of Inaticabtagene Autoleucel Injection (Experimental): Subjects who meet the enrollment conditions will receive intravenous infusion of CAR-T cells after lymphodepletion.
  Interventions: Drug: Inaticabtagene autoleucel Injection

INTERVENTIONS:
Drug: Inaticabtagene autoleucel Injection — Inaticabtagene autoleucel Injection, the autologous 2nd generation CD19-directed CAR-T cells, will be administered by vein. Before CAR-T infusion，patients will get a 3-4 days lymphodepletion therapy with fludarabine and cyclophosphamide.

SUMMARY:
This is a single-arm, open-label，phase I clinical study to evaluate the safety and tolerability of Inaticabtagene Autoleucel Injection in treatment of refractory systemic lupus erythematosus-related immune thrombocytopenia.

DETAILED DESCRIPTION:
This is a single arm, open-label, non-randomized, dose-escalation, phase I study to determine the safety and tolerability of Inaticabtagene Autoleucel Injection in treatment of refractory systemic lupus erythematosus-related immune thrombocytopenia and determine the Phase II Recommended Dose (RP2D). The study will have the following sequential phases: Screening, Pre-Treatment (Cell Product Preparation & Lymphodepleting Chemotherapy), Treatment and Follow-up, and Survival Follow-up. The total duration of the study is 2 years from Inaticabtagene Autoleucel Injection infusion.

ELIGIBILITY:
Inclusion Criteria:

1. Age range: 18-70 years (including 18 and 70 years), regardless of gender.
2. Clinically diagnosed with Refractory Systemic Lupus Erythematosus-related Immune Thrombocytopenia according to the revised criteria of ACR in 1997 or EULAR/ACR in 2019. At least two consecutive blood routine tests showing platelet counts <50×10^9/L; Peripheral blood smear microscopy showed no significant abnormalities in the morphology of blood cells; The morphological characteristics of bone marrow cells are consistent with immune thrombocytopenia. Treated at least 1 course of MP shock therapy or high-dose steroids, combined with one or more immunosuppressive agents (including biologics) for at least 3 months but not achieving partial remission, or the efficacy cannot be maintained during the steroid reduction process.
3. During the study period, the use of corticosteroids at a dose not exceeding 10mg prednisone or its equivalent, all immunosuppressants (excluding hydroxychloroquine) should be discontinued.
4. Women of childbearing potential must have a negative blood pregnancy test 7 days prior to trial conditioning therapy; any male and female patients of childbearing potential must agree to use an effective method of contraception throughout the study and for at least 2 year following infusion of CAR-T cells. Childbearing potential is biologically capable of bearing a living baby and sexually active. Female patients who were not of childbearing potential (ie, met at least 1 of the following criteria):

   * Hysterectomy or oophorectomy, or
   * Medically confirmed ovarian failure, or medically confirmed postmenopausal (cessation of menses for at least 12 consecutive months in the absence of pathological or physiological causes).
5. Adequate organ function according to the following criteria:

   * Aspartate aminotransferase (AST) ≤ 3 times of upper limit of normal (ULN);
   * Alanine aminotransferase (ALT) ≤ 3 times ULN;
   * Total serum bilirubin ≤ 2 times ULN unless the patient has documented Gilbert's syndrome; patients with Gilbert's syndrome who have bilirubin ≤ 3.0 times ULN and direct bilirubin ≤ 1.5 times ULN may be included;
   * Serum creatinine ≤ 1.5 times ULN, or creatinine clearance ≥ 60 mL/min (Cockcroft and Gault formula), Patients with lupus nephritis may relax the conditions appropriately according to the judgment of the investigator;
   * Must have minimal pulmonary reserve and oxygen saturation > 91% in a nonoxygenated state;
   * Lymphocyte count > 0.4 × 109/L.

Exclusion Criteria:

1. Severe active central nervous system (CNS) lupus, including seizures, psychosis, cerebrovascular accidents, or CNS vasculitis requiring therapeutic intervention within 60 days after baseline.
2. Dialysis patients or creatinine clearance rate less than 30mL/min.
3. Pregnancy or breastfeeding.
4. Merge active infections (such as sepsis, bacteremia, mycosis, uncontrolled lung infections, and active tuberculosis).
5. Hepatitis B surface antigen (HBsAg) and/or hepatitis B e antigen (HBeAg) are positive; Hepatitis B e antibody (HBe Ab) and/or hepatitis B core antibody (HBcAb) are positive, and the number of HBV-DNA copies is greater than the measurable lower limit; Hepatitis C (HCV) antibody positive; positive for human immunodeficiency virus (HIV) antibodies; positive for syphilis antibody (TP Ab);
6. Major surgery that was assessed as unsuitable by the investigators within 4 weeks before screening.
7. Patients with concurrent active malignancy within the past five years, those with a history of malignancy but cuired are eligible.
8. The patient's heart meets any of the following conditions:

   Left ventricular ejection fraction (LVEF) ≤ 45%; New York Heart Association (NYHA) Grade III or IV congestive heart failure or active heart disease; Severe arrhythmias that require treatment (excluding atrial fibrillation and paroxysmal supraventricular tachycardia); QTcB interval ≥ 450ms for males and ≥ 470ms for females (QTcB=QT/RR1/2); Have had myocardial infarction, bypass or stent surgery within the 6 months prior to the study; Other heart diseases that have been determined by researchers to be unsuitable for inclusion;
9. Patients with clinically significant pleural effusion during screening.
10. Patients vaccinated with a live vaccine within 6 weeks prior to screening.
11. Patients with deep vein thrombosis within 6 months prior to screening, or a history of pulmonary embolism.
12. Patients with a life expectancy of less than 6 months.
13. Patients participating in any other interventional clinical study or receiving treatment of an active investigational drug within 3 months or 5 half-lives for launched drugs prior to Inaticabtagene Autoleucel Injection infusion.
14. Patients with a history of epilepsy, cerebral ischemia/hemorrhage, cerebellar diseases, or other active central nervous system disorders;
15. Patients with hypersensitivity reactions to the components of Inaticabtagene Autoleucel Injection.
16. Patients previously received CAR-T cell therapy.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2025-03-01 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-related Adverse Events | Up to 28 days post-infusion
  Therapy-related adverse events (AE), including severe adverse events (SAE) and laboratory outliers with clinical significance, will be recorded and assessed according to the Common Terminology Criteria for Adverse Events (CTCAE, Version 5.0)
The safe dosage for a single infusion of Inaticabtagene Autoleucel Injection | Up to 28 days post-infusion
  The safe dosage for ITP patients will be evaluated by comprehensively assessing the Overall Response Rate (ORR) and the incidence of adverse events (AEs).

SECONDARY OUTCOMES:
Overall Remission Rate (ORR) | Up to 6 months post-infusion
  The proportion of subjects achieving CR or PR after treatment by Inaticabtagene Autoleucel Injection.CR is defined as platelet count ≥100×10^9/L. PR is defined as platelet count ≥30×10^9/L and at least doubling from baseline, without active bleeding.
Proportion of subjects who achieved disease remission (DORIS) | Up to 6 months post-infusion
  The proportion of subjects to meet the following 2 criteria: 1.Clinical lupus erythematosus disease activity index (SLEDAI)=0. 2.Physician global assessment (PGA) is less than 0.5 (standard score is 0-3 points) without considering serological testing and low dose corticosteroids with a dose of ≤ 5mg/d (taking prednisone as an example) permitted. Antimalarial drugs, stable dose immunosuppressants, including biologics are allowed to be used.
Proportion of subjects who achieved lupus hypoactivity state (LLDAS) | Up to 6 months post-infusion
  The proportion of subjects to meet the following 5 criteria:
  1. SLEDAI score ≤ 4, no activity of important organs, no hemolytic anemia or gastrointestinal activity;
  2. Compared with previous assessments, there is no new lupus activity;
  3. SELENA-SLEDAI physician overall assessment (PGA 0-3) ≤ 1 point;
  4. The current dose of prednisone is ≤ 7.5mg/d;
  5. Immunosuppressants and biologics with standard maintenance doses are well tolerated.
Improvement in systemic lupus erythematosus scores (SELENA-SLEDAI) | Up to 24 months post-infusion
  0 to 4 is basically no disease activity;5 to 9 is light activity;10 to 14 is moderate activity;≥15 is considered heavy activity.
Changes in MOS item short from health survey(SF-36) | Up to 24 months post-infusion
Changes in Primary Immune Thrombocytopenia Patient Assessment Questionnaire (ITP-PAQ) | Up to 24 months post-infusion
Changes in serological markers | Up to 24 months post-infusion
  Changes in IgG, IgM, IgA, IgE levels compared to baseline.
Changes in serological markers | Up to 24 months post-infusion
  Changes in SLE disease serological markers (anti ds-DNA antibody, anti nuclear antibody AG, complement C3, C4) levels compared to baseline.
Reduction of Combination therapy evaluation | Up to 24 months post-infusion
  The duration of the patient's cessation or reduction of the combination therapy dose, as well as the degree of reduction in the combination therapy compared to baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Mengtao Li, Dr., Principal Investigator — Peking Union Medical College
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China